CLINICAL TRIAL: NCT06746493
Title: Is it Important to Assess the Function of the Knee Joint After a Stroke
Brief Title: The Assessment of Knee Joints Function in People After Stroke
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Wareńczak-Pawlicka, Study Chair: Agnieszka Wareńczak-Pawlicka, PhD, Department of Rehabilitation and Physiotherapy Rehabilitation, Poznan University of Medical Sciences
Other Study IDs: 822/21
Record Dates: First submitted 2024-03-11; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: function of knee joint; physiotherapy; wireless sensors; functional tests
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke group: All patients from the stroke group were examined twice at the beginning and the end of this trial by a physical therapist. Patients participated in a rehabilitation program at the Neurological Rehabilitation Department between measurements.
  Interventions: Other: Rehabilitation
- Control group: The control group consisted of healthy subjects.

INTERVENTIONS:
Other: Rehabilitation — People after a stroke participated in a standard rehabilitation process carried out at the neurological rehabilitation department.
  Other Names: Physical rehabilitation
  Groups: Stroke group

SUMMARY:
The study aims to assess the function of knee joints in patients after stroke compared to healthy people and evaluate the impact of rehabilitation on the function of knee joints in people after stroke.

DETAILED DESCRIPTION:
Stroke patients were examined twice at the beginning of rehabilitation and after approximately 15 days of exercise. The control group (healthy participants) was assessed once. Wireless motion sensors connected to a mobile application were used to assess the kinematics of the knee joints. They were used to assess the range of motion in the knee joints (passive, active, active at maximum speed), proprioception (joint position sense tests), step-up test, step-down test, getting up and sitting on a chair, step and squat. Functional tests such as The Five Times Sit-to-Stand Test, Timed Up&Go, The Step Test, the 5m walking test, and the 30-s Chair Stand Test were carried out. The strength of the knee extensors and flexors was also assessed using the Leg Force Feedback device. Balance was assessed on a posturography platform by performing tests such as standing with eyes open and closed on a stable surface and standing with eyes open and closed on an unstable surface. The symmetry of lower limb loads in a standing position was also assessed.

ELIGIBILITY:
Inclusion criteria to the stroke group were as follows :

* the time from stroke: less than a year,
* age: between 35 and 65 years old,
* ability to stand independently for at least 5 minutes without an assistive device,
* ability to walk 5 m independently,
* ability to communicate and understand the tasks required in the study,
* a modified Ashworth scale spasticity score of 1+ or less in the affected knee (0: no resistance, 5: affected parts stiff in flexion or extension),
* muscle strength on the Manual Muscle Test of 3/4 or more in the affected knee,
* Barthel Index score 80 or more.

Exclusion criteria from the post-stroke group were as follows:

* age below 35 or over 65,
* sensorimotor aphasia,
* cognitive disorders that make it impossible to understand and obey commands,
* lack of active movement in the knee joint,
* Manual Muscle Test strength of the quadriceps muscles below 3,
* no ability to walk 5 meters,
* lack of informed consent to participate in the study,
* other neurological diseases (such as MS, Parkinson's disease, neuropathies),
* fractures in the lower limbs, which could affect the structure and function of the knee joint,
* previous operations on the lower limbs (including ACL reconstruction, knee arthroplasty or hip, osteotomy of the knee joint).
* vision disorders,
* unilateral spatial neglect syndrome.

The control group consisted of healthy volunteers with no prior history of trauma or neurological disease affecting the structure and function of the lower limb.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group comprised patients after stroke. The control group consisted of healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the passive and active range of motion of the knee joint using wireless motion sensors connected to a mobile application. | Baseline and after about 15 days of exercise.
  Measurement of the passive and active range of motion of the knee joint in degrees in lying position using wireless motion sensors connected to a mobile application.
Proprioception | Baseline and after about 15 days of exercise.
  Assessment of joint position sensation (3 different positions indicated) in degrees using wireless sensors.
Assessment of the active range of motion of the knee and hip joint during functional tasks | Baseline and after about 15 days of exercise.
  Measurement of the range of motion of the knee and hip joint using wireless motion sensors connected to a mobile application during functional tasks such as: step up, step down, squat, sitting on a chair and getting up from a chair and step forward.
Assessment of the maximum angle of varus and valgus at the knee joint during functional tasks | Baseline and after about 15 days of exercise.
  Measurement of the maximum angle of varus and valgus at the knee joint using wireless motion sensors connected to a mobile application during functional tasks such as: step up, step down, squat, sitting on a chair and getting up from a chair and step forward.
Assessment of the mean squared error at the knee joint during functional tasks | Baseline and after about 15 days of exercise.
  Measurement of the mean squared error using wireless motion sensors connected to a mobile application during active flexion and extension motion in the knee joint at maximum speed and functional tasks such as: step up, step down, squat, sitting on a chair and getting up from a chair and step forward.
Assessment of the speed of movement in the knee joint during functional tasks | Baseline and after about 15 days of exercise.
  Measurement of the speed of movement in the knee joint during active flexion and extension motion in the knee joint at maximum speed and functional tasks such as: squat and sitting on a chair and getting up from a chair.
Step test | Baseline and after about 15 days of exercise.
  Assessment of the number of repetitions.
The Five Times Sit-to-Stand Test | Baseline and after about 15 days of exercise.
  Assessment of task completion time.
Timed Up&Go Test | Baseline and after about 15 days of exercise.
  Assessment of task completion time.
30-s Chair Stand Test | Baseline and after about 15 days of exercise.
  Assessment of the number of repetitions.
5m walking test | Baseline and after about 15 days of exercise.
  Assessment of task completion time.
Assessment of isometric muscle strength of knee flexors and extensors using Leg Force Feedback device. | Baseline and after about 15 days of exercise.
  Measurement of the maximal voluntary isometric contraction torque of the knee extensor and flexor muscle groups in Newton-meter.
Symmetry | Baseline and after about 15 days of exercise.
  Assessment of the load on the lower limbs while standing in percentage.

SECONDARY OUTCOMES:
Assessment of the center of pressure path length when measuring on a balance platform | Baseline and after about 15 days of exercise.
  Measurement of parameter such as total path length (cm). A test was performed in four conditions: standing with eyes open and closed on a stable surface and standing with eyes open and closed on an unstable surface.
Assessment of the center of pressure velocity when measuring on a balance platform | Baseline and after about 15 days of exercise.
  Assessment of parameter such as average speed (cm/s). A test was performed in four conditions: standing with eyes open and closed on a stable surface and standing with eyes open and closed on an unstable surface.
Balance | Baseline and after about 15 days of exercise.
  The test was performed in four conditions: standing with eyes open and closed on a stable surface and standing with eyes open and closed on an unstable surface. The results were obtained in percentage values and compared to the normative results from the system.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Wareńczak-Pawlicka, PhD, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
The data is available in the form of an anonymized CSV sheet.